CLINICAL TRIAL: NCT02027662
Title: Study to Investigate Efficacy and Safety Equivalence of OsvaRen® Tablets and OsvaRen® Granules
Brief Title: Therapeutic Equivalence of OsvaRen® Tablets and OsvaRen® Granules
Acronym: OsvaRenNEW
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Fresenius Medical Care Deutschland GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: RP-OSV-02-D
Record Dates: First submitted 2013-12-20; First posted 2014-01-06 (Estimated); Last update posted 2015-06-10 (Estimated); Status verified 2015-06

CONDITIONS: Hyperphosphatemia; Chronic Kidney Disease
MeSH Terms: conditions — Hyperphosphatemia; Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Osvaren Granules (Experimental): Osvaren Granules
  Interventions: Drug: Osvaren Granules
- Osvaren film-coated tablets (Active Comparator): Osvaren film-coated tablets
  Interventions: Drug: Osvaren film-coated tablets

INTERVENTIONS:
Drug: Osvaren Granules
  Arms: Osvaren Granules
Drug: Osvaren film-coated tablets
  Arms: Osvaren film-coated tablets

SUMMARY:
Phosphate binders are crucial to the control of elevated phosphate levels in patients with chronic kidney disease. With the new formulation of granules the pill burden of patients is sought to be reduced.

This study is about efficacy and safety of the new drug formulation and compares it to the "old" formulation which are film-coated tablets.

DETAILED DESCRIPTION:
The study is aimed at demonstrating the therapeutic equivalence of both products, i.e. granules versus tablets.

Secondary objectives are: Comparing both preparations with regard to the number of patients reaching serum phosphate levels < 1.76 mmol/L and the difference in serum phosphate levels between the first and last visit under each treatment. Furthermore, it is the aim of this study to evaluate the safety profile of OsvaRen® granules in comparison to OsvaRen® tablets. Especially serum calcium, magnesium, and PTH are of interest.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent form is obtained prior to starting the screening visit
* Male and female patients 18-80 years of age with dialysis dependent renal failure (CKD 5D)
* Patients have been on 3x/week in-centre renal replacement therapy for at least 2 months on either low-flux or high-flux HD or OL-

  /HDF
* Prescribed haemodialysis session duration is ≥ 4 hours
* spKt/V ≥ 1.20 according to last in-centre measurement prior the study enrolment
* Patients have been on OsvaRen® tablets for at least 12 weeks as sole phosphate binder and the titration phase has been completed according to physician´s discretion
* Patients are able to take the study medication as prescribed particularly OsvaRen® stickpacks
* Patients are willing to stop any calcium, magnesium or vitamin D containing supplements
* Patients are willing to maintain their typical diet with regards to phosphate uptake for the time of the study
* Patients are willing to comply with the study protocol

Exclusion criteria

* Pregnant women (by blood ß-hCG pregnancy test) or women breast-feeding or unwilling to use contraceptive measures during the entire course of the study or
* Patients with a life expectancy shorter than the planned duration of the study or
* Patients with any acute or chronic severe disease potentially interfering with study outcomes or
* Patients with PTH levels > 800 ng/l or
* Patients who participated in an interventional clinical study during the preceding 30 days or
* Patients suffering from any other, not mentioned condition which could interfere with the patient's ability to comply with the study or
* Patients who previously participated in the same study are excluded from the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2014-01; Primary Completion 2015-04 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Non-inferiority of phosphate control by granules versus tablets. Serum phosphate levels will be measured for the primary outcome. | After 4 weeks of treatment time

SECONDARY OUTCOMES:
Number of patients reaching serum phosphate levels < 1.76 mmol/L. this study to evaluate the safety profile of OsvaRen® granules. in comparison to OsvaRen® tablets. Especially serum calcium, magnesium, and PTH are of interest. | Between the first and last visit under each treatment i.e. 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jürgen Floege, MD, Principal Investigator — University Aachen
Locations (11):
- Germany (11):
  - Georg-Haas-Dialysezentrum der PHV, Giessen, Hesse
  - RWTH University Hospital, Dpt for Nephrology, Aachen, North Rhine-Westphalia
  - Nephro-Studien GbR am Klinikum Erfurt, Erfurt
  - Dialysezentrum, Flensburg
  - Nephrocare Hamburg-Barmbek GmbH, Hamburg
  - Dialysezentrum, Hanover
  - Dialysezentrum, Kiel
  - Dialysezentrum, Magdeburg
  - Dialysezentrum, Minden
  - Dialysezentrum, Solingen
  - Dialysezentrum, Velbert

REFERENCES:
- [Derived] Natale P, Green SC, Ruospo M, Craig JC, Vecchio M, Elder GJ, Strippoli GF. Phosphate binders for preventing and treating chronic kidney disease-mineral and bone disorder (CKD-MBD). Cochrane Database Syst Rev. 2025 Jun 27;6(6):CD006023. doi: 10.1002/14651858.CD006023.pub4. PMID 40576086